CLINICAL TRIAL: NCT06754579
Title: Effect of High-Volume Upper Extremity Exercises on Physical and Cognitive Performance in Sedentary Adults
Brief Title: Impact of High-Volume Upper Limb Training on Physical and Cognitive Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Fatma Kübra ÇEKOK, Asst.prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Behavior
Keywords: upper limb; reaction time; pyhsical performance; cognitive performance
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled study
Who Masked: Participant
Masking Description: Study participants are unaware of their assigned group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Volume Upper Extremity Exercises Training (Experimental): The High volume upper extremity protocol consists of a 5-min warm-up at 60%-70% of max HR using an arm ergometer, followed by four 4-min work sessions reaching 90%-95% of max W, followed by a 3-min active recovery period at 60% max W. The exercise session is terminated by a 5-min cool-down at 60%-70% max W. The total exercise duration will be 35 minutes.
  Interventions: Other: High-Volume Upper Extremity Exercises Training
- Low Volume Upper Extremity Exercises Training (Experimental): Low volume upper extremity exercise training will be applied using an arm ergometer consisting of a 5-minute warm-up at 40% of max W, followed by 25 minutes of active training at 60-70% of max W and a 5-minute cool-down at 40% of max.
  Interventions: Other: Low Volume Upper Extremity Exercises Training

INTERVENTIONS:
Other: High-Volume Upper Extremity Exercises Training — The group will be trained 3 days a week for a total of 8 weeks.
  Arms: High-Volume Upper Extremity Exercises Training
Other: Low Volume Upper Extremity Exercises Training — The group will be trained 3 days a week for a total of 8 weeks.
  Arms: Low Volume Upper Extremity Exercises Training

SUMMARY:
Engaging in regular and appropriately structured physical activities is a critical component of an individual's lifestyle and represents a lifelong habit essential for promoting overall well-being. Research increasingly emphasizes the significance of such activities, particularly in the prevention and management of various health conditions (Martin, Richardson, Weiller, & Jackson, 2004).A sedentary lifestyle is considered one of the most serious health issues faced by individuals in the modern world.Previous research has established high-intensity interval training (HIIT) as an effective method for enhancing cardiovascular health, sparking interest in the relationship between exercise intensity and cognitive function. Most studies to date have focused on treadmill and lower extremity ergometer exercises; however, evidence regarding the efficacy of high-volume upper extremity exercises in improving physical and cognitive performance among sedentary adults remains limited and inconsistent. Upper extremity motor function has been proposed as a potential biomarker for cognitive impairment and may contribute to distinguishing healthy aging trajectories. This study aims to compare the effects of high-volume and low-volume upper extremity exercise in sedentary adults, testing the hypothesis that one exercise regimen may be superior in enhancing both physical and cognitive performance, as well as cognitive function.

DETAILED DESCRIPTION:
Engaging in regular, well-structured physical activities is a cornerstone of a healthy lifestyle and constitutes a lifelong habit essential for sustaining overall health and well-being. Such activities have been increasingly recognized for their vital role in preventing and managing a wide range of health conditions, emphasizing their importance for both physical and mental health (Martin, Richardson, Weiller, & Jackson, 2004). Conversely, a sedentary lifestyle has emerged as one of the most pressing public health challenges of the modern era, contributing significantly to the global burden of disease and highlighting the need for effective intervention strategies.

Among these strategies, high-intensity interval training (HIIT) has gained widespread attention for its efficacy in improving cardiovascular health. This has, in turn, sparked growing interest in understanding the broader impact of exercise intensity, particularly its effects on cognitive function. However, much of the existing research has concentrated on lower extremity exercises, such as those performed on treadmills or ergometers, leaving a significant gap in the understanding of the benefits of upper extremity exercises. The role of high-volume upper extremity exercise in enhancing both physical and cognitive performance remains underexplored, with current evidence presenting inconsistent and conflicting findings.

Notably, upper extremity motor function has been identified as a promising biomarker for cognitive impairment. Its assessment may provide critical insights into distinguishing healthy aging trajectories from pathological cognitive decline. This connection underscores the potential importance of upper extremity exercises as a tool for both physical and cognitive health maintenance in sedentary populations.

The present study aims to address these gaps by comparing the effects of high-volume and low-volume upper extremity exercise regimens on sedentary adults. Specifically, the research seeks to test the hypothesis that one of these exercise modalities may offer superior benefits in enhancing physical performance, cognitive performance, and overall cognitive function. By investigating these relationships, the study aims to contribute to the growing body of evidence on exercise-based interventions, offering novel insights into strategies for optimizing health outcomes in sedentary individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-50 years.
* Defined as engaging in less than 150 minutes of moderate-intensity physical activity per week

Exclusion Criteria:

* diagnosis of neurological, cardiovascular, musculoskeletal, or other systemic diseases that may affect physical activity or exercise capacity.
* diagnosed cognitive impairments or psychiatric disorders that could interfere with test participation.
* acute injuries or surgeries within the past six months that could restrict movement or participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Short Form (IFQQ-SF) | eight weeks
  International Physical Activity Questionnaire-Short Form (IFQQ-SF): UFQ-SF was developed by Craig and colleagues to determine the physical activity levels of individuals between the ages of 15-65. The short form is recommended more because the long form is boring and repetitive, so the "last 7 days" short form was used in our study. The short form (7 questions) provides information on time spent in sitting, walking, moderate-intensity and vigorous activities. The total score is expressed as one MET-min/week and is obtained by multiplying the number of days and minutes of walking, moderate-intensity and vigorous activity and the MET score.

SECONDARY OUTCOMES:
Maximal Arm Exercise Capacity | Eight weeks
  The arm ergometer test is a widely used method to evaluate maximal arm exercise capacity, requiring the involvement of chest, back, hip, and leg muscles for body stabilization. This is particularly important as the test primarily targets a smaller muscle mass compared to bicycle ergometer testing. For this study, the Monark 881E Rehab Trainer (MONARK 881E, Monark, Varberg, Sweden) arm ergometer will be employed.
Stroop Test | Eight weeks
  The Stroop Test utilized in this study is based on the Istanbul Medical Faculty (Çapa) Neuropsychology Laboratory adaptation of the Stroop Test form originally developed by Weintraub (2000). Participants are instructed to name the colors of the small rectangles (red, blue, green) as quickly as possible, moving from left to right. This stage is used to identify any visual or color perception impairments, such as color blindness. If such deficiencies are detected, the test is discontinued.Stroop B (word reading): Participants are asked to read aloud the printed color names (red, blue, green) that are written in incompatible ink colors as quickly as possible. Stroop C (Color-Word Interference).
Reaction Time | Eight weeks
  The auditory and visual reaction times of sedentary individuals will be assessed using the Newtest 1000™ device (OY, Oulu, Finland). This device is capable of delivering three types of stimuli and consists of two primary components designed for precise reaction time measurements.Following the familiarization trial, three measurements will be conducted for each type of stimulus (auditory and visual), and the reaction times will be recorded in milliseconds. This protocol ensures the reliability of the data and accounts for variability in individual performance.
Hole Type Steadiness Tester | Eight weeks
  The participant will be asked to hold a metal tipped pencil with his dominant hand for 15 seconds in the 9 holes that are gradually decreasing in size without touching the edges. The purpose of the test will be to analyze the stability of the hand, exercise, smoking, alcohol intake, psychomotor speed, exercise and fatigue. Errors that occur when the participant touches the hole area will be recorded digitally. The test will be repeated 3 times on average and the result value will be calculated.
Postural Sway Assessment | Eight weeks
  Postural sway was assessed using the GYKO body sway device (Microgait, Italy), a validated tool that measures sway along two axes: mediolateral and anteroposterior (Jaworski et al., 2020). During the assessment, participants were instructed to stand in an upright posture with their feet positioned 10 cm apart and to maintain this posture for a duration of 30 seconds.
  Each participant underwent two trials under different visual conditions: eyes open and eyes closed. The mediolateral and anteroposterior sway distances were recorded for each trial. Data were automatically captured and stored in the accompanying computer software for subsequent analysis. This protocol ensures a reliable evaluation of postural control and stability under varying sensory conditions.
Upper Extremity Muscle Strength Assessment | Eight weeks
  MicroFET 2 muscle strength is a usable method for measuring muscle strength (Malliopoulos & Thevenon, 2002). Muscle strength is defined as the highest (maximal) voluntary contraction that the subject can perform under specific test conditions. The individual performed the highest voluntary contraction 3 times for each test. The individual increases his strength for 2 seconds and maintains it at the highest level for 3 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Kübra Çekok, Tarsus, Mersi̇n, Turkey (Türkiye)